CLINICAL TRIAL: NCT02049554
Title: Preconception Women's Health in Pediatric Practice Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Zanvyl and Isabelle Krieger Fund (Other); Abell Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NA_00084255
Record Dates: First submitted 2014-01-24; First posted 2014-01-30 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Preconception Care; Women's Health
Keywords: preconception care; women's health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention)
- Preconception Care Screener Group (Experimental): Women's Health Screener and Clinician discussion
  Interventions: Other: Preconception Care Screener

INTERVENTIONS:
Other: Preconception Care Screener
  Arms: Preconception Care Screener Group

SUMMARY:
The aims of the intervention are:

1. Assess the feasibility and effectiveness of preconception health care initiated by pediatric clinicians on outcomes including women's access to primary care and contraceptive services; contraception and rapid repeat pregnancy rate and interpregnancy interval; and women's immunization rate, control of chronic illnesses, nutritional status, smoking and substance use, mental health and violence exposure; child and family health.
2. Assess the cost-effectiveness of preconception health care initiated in pediatric practices.

The investigators will evaluate these outcomes with a clinic based trial comparing usual care to preconception care intervention.

ELIGIBILITY:
Inclusion Criteria:

Mothers with children ages 0 to 12 months presenting with their child for care at a participating pediatric office.

Exclusion Criteria:

-

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 415 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Receipt of preconception care | 6 months
Receipt of Preconception Care | 12 months

SECONDARY OUTCOMES:
Use of Highly Effective Contraception | 6 months
Use of Highly Effective Contraception | 12 months
Attendance at Preventive Health Care Visit | 6 months
Attendance at Preventive Health Care Visit | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Harriet Lane Clinic, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Chilukuri N, Cheng TL, Psoter KJ, Mistry KB, Connor KA, Levy DJ, Upadhya KK. Effectiveness of a Pediatric Primary Care Intervention to Increase Maternal Folate Use: Results from a Cluster Randomized Controlled Trial. J Pediatr. 2018 Jan;192:247-252.e1. doi: 10.1016/j.jpeds.2017.09.020. PMID 29246348